CLINICAL TRIAL: NCT02378870
Title: A Randomised, Double-blind, Placebo-controlled Multicentre Phase II Study to Evaluate Efficacy and Tolerability of ODX (Osteodex) in Metastatic Castration Resistant Prostate Cancer (CRPC)
Brief Title: A Phase IIb Study to Evaluate Efficacy and Tolerability of ODX (Osteodex) in Metastatic CRPC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor patient recruitment
Sponsor: DexTech Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ODX-002
Record Dates: First submitted 2014-11-17; First posted 2015-03-04 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer Metastatic
Keywords: CRPC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A:Osteodex (Experimental): 3.0 mg/kg bodyweight solution for infusion
  Interventions: Drug: Osteodex
- B: Placebo (Placebo Comparator): NaCl 0.9% solution for infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Osteodex — Osteodex 3.0 mg/kg given every two week, maximum 13 times.
  Other Names: ODX
  Arms: A:Osteodex
Drug: Placebo
  Arms: B: Placebo

SUMMARY:
This phase IIb study is a randomized, double-blind, placebo-controlled multi-center study evaluating efficacy and tolerability of Osteodex of patients with metastatic castration resistant prostate cancer (CRPC). Osteodex is a poly-bisphosphonate containing three known substances; dextran, alendronate and guanidine.

The objective of the study is to evaluate the relative change of response markers to bone metabolism (B-ALP and S-P1NP) The following objectives will also be evaluated: overall survival, PSA response, other response markers related to bone metabolism (S-CTX and osteocalcin), safety, tolerability, pain and quality of life.

DETAILED DESCRIPTION:
Males, diagnosed with CRPC, who fulfil the inclusion criteria and does not have any exclusion criteria, will be asked to participate in the study. The subject will be informed orally and in writing about the study procedures and give written informed consent, prior to study start. At the screening visit the following examinations are performed: Physical examination, medical history and concomitant medication. Heart rate, blood pressure, weight, height, body temperature and respiratory rate are measured. Blood samples are drawn and urine sample is collected. ECG is recorded. Bone scan and PET-CT are also performed. At the next visit, baseline, the subject is examined physically and heart rate, blood pressure, weight, body temperature and respiratory rate are measured, ECG is recorded, blood samples drawn and urine sample collected. FACT-P and EQ-5D-5L questionnaire are filled out by the subject. Adverse events and concomitant medication is documented and the first dose of the investigational product is given.

The subject is surveyed for 3 hours at the hospital.

The duration of the study for the individual subject will be approximately 30 weeks from screening to the follow-up visit 2 weeks after the last dose. Each subject will receive at least 7 doses and maximum 13 doses of investigational product.

A Data Monitoring Committee (DMC) will be designated and will be responsible to monitor/review all study related safety data. After review of safety data the DMC will provide recommendation as to whether the dose escalation can proceed as planned according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent form.
2. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate.
3. Failing or not tolerating docetaxel therapy or for other reasons not suitable for such therapy and failing subsequent therapy with abiraterone and/or enzalutamide.
4. Evidence of metastatic disease from bone scan (bone lesions) or other imaging modality.
5. Evidence of PSA progression in two consecutive determinations at minimum 1 week interval.
6. Castrate level of serum testosterone ≤1.7 nmol/L
7. Performance status ECOG 0-2
8. Laboratory requirements: Haematology: Neutrophils ≥ 1.5 x 109/l Hemoglobin ≥ 90 g/l Platelets ≥ 100 x 109/l Hepatic function: Total S-bilirubin ≤ 1.5 times the upper limit of normal (ULN) AST (SGOT) / ALT (SGPT) ≤ 2.5 times ULN Renal function: S-creatinine ≤ 1.5 times the upper limit of normal (ULN) Electrolytes: S-sodium, S-potassium, S-calcium (S-albumin corrected), S-phosphate, S-magnesium, all within normal ranges.
9. No evidence (≤ 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).
10. Able to adhere to the study visit schedule and other protocol requirements.
11. Life expectancy ≥6 months

Exclusion Criteria:

1. Concurrent use of other anti-cancer agents or treatments, with the following exception: a stable dose of LHRH agonist/antagonist or polyestradiol phosphate bicalutamide. Washout period bicalutamide 6 weeks; after flutamide 4 weeks; abiraterone / enzalutamide 6 weeks.
2. Any treatment modalities involving chemotherapy, radiation or major surgery within 4 weeks prior to treatment in this study.
3. Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to start of study treatment.
4. Any condition, including the presence of laboratory abnormalities, which confounds the ability to interpret data from the study or places the patient at unacceptable risk if he participates in the study.
5. Plasma glucose level ≥7 mmol/l (or >120 mg/dl) at screening.
6. Known brain metastases.
7. Dental surgery (dental extraction), periodontal disease, local trauma including poorly fitting dentures within 6 months prior to the first dose of study drug.
8. Treatment with bisphosphonates within 4 weeks prior to first dose of study medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Relative change in response markers related to bone metabolism (B-ALP and S-P1NP) | Baseline and 24 weeks of treatment

SECONDARY OUTCOMES:
Relative change in response markers related to bone metabolism (B-ALP and S-P1NP) | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22 weeks of treatment and at 2 weeks post-treatment.
Relative change in response markers related to bone metabolism (S-CTX and osteocalcin) | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment.
PSA response | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment.
Overall survival | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment. Long-term follow-up will be conducted every 3rd month, up to 12 months.
  Life expectancy for participating subjects ≥ 6 months
Pain | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment.
  FACT-P questionnaire
Analgesic consumption | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment. Long-term follow-up will be conducted every 3rd month, up to 12 months.
  Life expectancy for participating subjects ≥ 6 months
Changes in tumor cell metabolism measured | Baseline, 12 and 24 weeks of treatment
  PET-CT
Changes in bone metastasis | Baseline, 12 and 24 weeks of treatment
  Bone scan
Incidence, causality and intensity of AEs | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment. Long-term follow-up will be conducted every 3rd month, up to 12 months
  Life expectancy for participating subjects ≥ 6 months
Dose and duration of medications required for the treatment of AEs | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and at 2 weeks post-treatment. Long-term follow-up will be conducted every 3rd month, up to 12 months.
Change from baseline in Quality of life | Baseline and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 weeks of treatment and 2 weeks post-treatment.
  EQ-5D-5L questionnaire, FACT-P questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Thellenberg-Karlsson, MD, PhD., Principal Investigator — Oncology Department, Norrland University Hospital (NUS) Umeå Sweden; Claes Nyman, MD, PhD., Principal Investigator — Urology Clinic, Stockholm South General Hospital (SÖS) Stockholm Sweden; Henriette Lindberg, MD, PhD., Principal Investigator — Oncology Department, Herlev Hospital, Copenhagen Denmark; Anders R Holmberg, CEO, Study Director — DexTech Medical AB
Locations (1):
- Oncology clinic, Norrlands Universitetssjukhus, Umeå, Umeå, Sweden